CLINICAL TRIAL: NCT04243174
Title: The Use of Mobile Phone Messaging as a Behavioural Intervention to Increase Physical Activity in Adults With T2DM in Saudi Arabia
Brief Title: The Use of Short SMS Messaging With Type 2 Diabetes (T2DM)
Acronym: mHealth
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Nottingham (Other)
Responsible Party: Principal Investigator, Holly Blake, Associate Professor, University of Nottingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 10
Record Dates: First submitted 2019-11-19; First posted 2020-01-28 (Actual); Last update posted 2021-08-27 (Actual); Status verified 2021-08

CONDITIONS: Type 2 Diabetes; Physical Exercise
MeSH Terms: conditions — Diabetes Mellitus, Type 2; Motor Activity

STUDY DESIGN:
Intervention Model Description: Single Group where they start receiving SMS messages about the importance of physical activity and its benefits on T2DM.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SMS Messages (Other): Patients with type 2 diabetes will be recruited and will start receiving short SMS messages about physical activity, encouraging them to be more active and help them to build a healthy life style routine.
  Interventions: Behavioral: SMS Messaging

INTERVENTIONS:
Behavioral: SMS Messaging — Patients with type 2 diabetes will be recruited and will start receiving short SMS messages about physical activity, encouraging them to be more active and help them to build a healthy life style routine.

SUMMARY:
Physical activity (PA) can play a vital and an independent role in type 2 diabetes (T2DM) management care. Health research studies have shown evidence that PA can improve glycaemic control and glucose levels. PA is first line of self-care management recommended to patients with T2DM and most patients fail to perform the regular PA. It is always important for health providers to find better methods in encouraging and incentivizing PA in T2DM patients. Mobile phone messaging-based interventions have been shown to strengthen the delivery of health information and self-care management programs.

DETAILED DESCRIPTION:
Studies have employed this as a tool for promoting T2DM self-care management interventions such as physical activity, glucose monitoring, medication adherence and nutrition. Despite the increasing number of these interventions globally, the effectiveness of mobile phone messaging-based interventions in Saudi Arabia context remains inconclusive and inconsistent. There is limited research conducted in this region. Therefore, there is a need for more studies to show evidence to ascertain the effectiveness of using mobile phone messaging to promote PA in T2DM patients in the context of Saudi Arabia.

ELIGIBILITY:
Inclusion Criteria:

* Clinician diagnosis of T2DM.
* Over 18 years of age.
* Possession of a cell phone with text messaging capability.
* Ability to read and understand Arabic.

Exclusion Criteria:

* Treatment with insulin adjustment
* Unable to understand the study requirements or give informed consent.
* Visual impairment.
* Any diabetes-related complications such as neuropathy or retinopathy that preclude ability to increase PA.
* Clinician concern (physicians will be asked to confirm whether eligible participants can be medically capable of performing PA at the recommended level advised by National Institute for Health and Care Excellence (NICE, 2013).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 57 (Actual)
Dates: Start 2020-01-23 (Actual); Primary Completion 2020-03-01 (Actual); Study Completion 2020-03-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of mobile phone text messaging intervention for people with T2DM: Number of Participants recruited, completed the study, dropped out | Six weeks
  Number of Participants recruited, completed the study, dropped out.

SECONDARY OUTCOMES:
Acceptability of mobile phone text messaging intervention for people with T2DM: Qualitative interviews | Six weeks
  Qualitative interviews will be undertaken with study participants and healthcare professionals (HCPs) to explore: satisfaction with the intervention; barriers and facilitators of the intervention; perceived impact of the intervention, and potential changes and necessary improvements.
Clinical measurements pre and after the intervention | 3 months
  Is glycated haemoglobin (HbA1c) sensitive to change when using SMS text messaging for physical activity promotion in the care of T2DM
Clinical measurements pre and after the intervention | 3 months
  Is the body mass index (BMI) in kg/m^2 sensitive to change when using SMS text messaging for physical activity promotion in the care of T2DM
Behaviour change outcome | Six weeks
  Is self-efficacy for physical activity (SEPA) questionnaire sensitive to change when using SMS text messaging for physical activity promotion in the care of T2DM. The total score is calculated by finding the sum of the all items. The total score ranges between 10 and 40, with a higher score indicating more self-efficacy.
Self-report questionnaire (International Physical Activity Questionnaire - IPAQ) | Six weeks
  To compare levels of physical activity (PA) before and after an intervention, IPAQ is used to assess moderate-to-vigorous physical activity in adult people. Categorical Score- three levels of physical activity are proposed:
  1. Low
     • No activity is reported.
  2. Moderate
     * More days of vigorous activity of at least 20 minutes per day.
       3. High
     * Vigorous-intensity activity on at least 3 days and accumulating at least 1500MET-minutes/week.

CONTACTS AND LOCATIONS:
Overall Officials: Dr.Holly Blake, PhD, Principal Investigator — University of Nottingham
Locations (1):
- King Fahd Medical City, Riyadh, Saudi Arabia

IPD SHARING:
Plan to Share IPD: Yes
After the study has been conducted and completed.
Supporting Information: Study Protocol
Time Frame: 01-06-2020